CLINICAL TRIAL: NCT01910441
Title: A Comparative Study to Assess the Effect of Vildagliptin Versus Glimepiride on Glucose Variability in Type 2 Diabetic Patients Uncontrolled on Metformin Alone
Brief Title: Comparison of Vildagliptin vs. Glimepiride on Glucose Variability in Metformin Uncontrolled Type 2 Diabetic Patients
Acronym: VARIABLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to the unavailability of Continuous Glucose Monitoring sensors (CGMS) which were required to assess the primary end-point.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AIN03
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Vildagliptin plus metformin (Experimental): Participants received Vildagliptin 50 mg twice daily as an add-on to metformin (1000-1500mg daily).
  Interventions: Drug: Vildagliptin; Drug: Metformin
- Group B: Glimepiride plus metformin (Active Comparator): Participants received Glimepiride 1-6 mg once daily as an add-on to metformin (1000-1500mg daily).
  Interventions: Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50 mg twice daily
  Arms: Group A: Vildagliptin plus metformin
Drug: Glimepiride — Glimepiride 1-6 mg once daily
  Arms: Group B: Glimepiride plus metformin
Drug: Metformin — Metformin (1000-1500 mg daily)

SUMMARY:
Compare the effect of Vildagliptin plus Metformin versus Glimepiride plus Metformin on glucose variability in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given written informed consent to participate in the study.
2. Type 2 Diabetes Mellitus patients either Male or female from 18 - 75 years of age (both inclusive).
3. Patients who are uncontrolled on metformin monotherapy for at least past 4 weeks (1000-1500 mg daily and HbA1c > 7.5 - 9%).
4. Patients with HbA1C levels within the range > 7.5% - 9%. (If a past value is available within the last 12 weeks, it would be considered acceptable provided it was obtained after at least 4 weeks of metformin therapy 1000-1500 mg daily).

Exclusion Criteria:

1. Age > 75 years ; BMI <22 or >40 kg/m2
2. Patients who are on Insulin therapy at the time of study entry.
3. Type 1 Diabetes Mellitus patients.
4. Patients with severe renal (creatinine clearance < 50 ml/min) or hepatic impairment (including pre-treatment ALT or AST > 3 x ULN).

   Creatinine clearance will be estimated from serum creatinine using Cockcroft-Gault formula (Cockcroft and Gault, 1976)
5. Patients with contraindications as mentioned in the Summary of Product Characteristics (SPCs) for vildagliptin, metformin, glimepiride, vildagliptin plus metformin and glimiperide plus metformin.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: Glimepiride Plus Metformin: Participants received Vildagliptin 50 mg twice daily as an add-on to metformin (1000-1500mg daily).
Period: Overall Study
Arm/Group | Group A: Vildagliptin Plus Metformin | Group B: Glimepiride Plus Metformin
Started | 48 | 47
Completed | 41 | 37
Not Completed | 7 | 10
Not completed — Sponsor decision | 0 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Vildagliptin Plus Metformin | Group B: Glimepiride Plus Metformin | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (11.86) | 52.1 (9.29) | 50.9 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 36
  Male | 26 | 33 | 59

OUTCOME MEASURES:

1. Primary Outcome: Mean Amplitude of Glycemic Excursions (MAGE)
Time Frame: 16 weeks
Population: The study was prematurely terminated due to the unavailability of CGMS required for the assessment of the primary end point. The non-availability of CGMS severely affected participant recruitment. The primary outcome was not analyzed.
Arm/Group | Group A: Vildagliptin Plus Metformin | Group B: Glimepiride Plus Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A: Vildagliptin Plus Metformin | Group B: Glimepiride Plus Metformin
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/47
Other Adverse Events (participants affected / at risk) | 4/48 | 1/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Vildagliptin Plus Metformin (N=48) | Group B: Glimepiride Plus Metformin (N=47)
HEADACHE (Nervous system disorders) | 0 | 1
RESTLESSNESS (Psychiatric disorders) | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Vildagliptin Plus Metformin (N=48) | Group B: Glimepiride Plus Metformin (N=47)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.